CLINICAL TRIAL: NCT02331680
Title: A Phase 2, Multicenter, Placebo-controlled, Double-blind, Randomized, Parallel-group Trial to Investigate the Efficacy and Safety of Orally Administered Tolvaptan (OPC-41061) in Patients With Chronic Renal Failure Undergoing Hemodialysis or Hemodiafiltration
Brief Title: A Trial to Investigate the Efficacy and Safety of Orally Administered Tolvaptan (OPC-41061) in Patients With Chronic Renal Failure Undergoing Hemodialysis or Hemodiafiltration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-13-003; JapicCTI-142756 (Other: Japic)
Record Dates: First submitted 2014-12-23; First posted 2015-01-06 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Renal Failure
Keywords: Undergoing Hemodialysis; Undergoing Hemodiafiltration
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPC-41061 15mg/day (Experimental): Will be orally administered once daily after breakfast on all days on which subjects do not undergo dialysis. OPC-41061 at 15 mg/day will be administered for 24 week.
  Interventions: Drug: OPC-41061
- OPC-41061 30mg/day (Experimental): Will be orally administered once daily after breakfast on all days on which subjects do not undergo dialysis. OPC-41061 at 15 mg/day will be administered for 1 week and then OPC-41061 30 mg/day for 23 weeks
  Interventions: Drug: OPC-41061
- Placebo (Placebo Comparator): Will be orally administered once daily after breakfast on all days on which subjects do not undergo dialysis. Placebo will be administered for 24 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-41061
  Other Names: Tolvaptan
  Arms: OPC-41061 15mg/day
Drug: OPC-41061
  Other Names: Tolvaptan
  Arms: OPC-41061 30mg/day
Drug: Placebo
  Other Names: Blank Tablet
  Arms: Placebo

SUMMARY:
This is a study to investigate the efficacy and safety of OPC-41061 by 24-week oral administration of OPC-41061 at 15-mg or 30-mg or placebo in patients with chronic renal failure who are undergoing hemodialysis or hemodiafiltration and who have daily urine volume of at least 500 mL/day.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure requiring hemodialysis or hemodiafiltration 3 times a week
* Daily urine volume of ≥ 500 mL/day
* Male or female patients age 20 to 80 years, inclusive
* Use of one of the specified contraceptive methods until 4 weeks after final IMP administration
* Capable of providing their own written informed consent prior to any trial-related procedures being performed

Exclusion Criteria:

* Patients with a complication of urinary impairment due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
* Patients with NYHA class IV heart failure
* Patients with impaired hepatic function(chronic hepatitis, drug-induced liver injury)
* Patients with serious ischemic heart disease who are judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial
* Patients with serious arrhythmia who are judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial
* Patients with serious secondary hyperparathyroidism(intact parathyroid hormone > 500 pg/mL)
* Patients who are concomitantly undergoing peritoneal dialysis
* Patients with a history of cerebrovascular disease or coronary artery disease within 4 weeks prior to informed consent, a history of hypersensitivity to any ingredient of tolvaptan or benzazepine derivatives such as mozavaptan hydrochloride or a history of impaired hepatic function(chronic hepatitis, drug-induced liver injury)
* Patients with any of the following abnormal laboratory values: hemoglobin < 8.0 g/dL, total bilirubin > 3.0 mg/dL, ALT (GPT) or AST (GOT) > 2 times the upper limit of the reference range, serum sodium > upper limit of the reference range, serum sodium < 125 mEq/L, or serum potassium > 6.0 mEq/L
* Patients who are unable to sense thirst or who have difficulty with fluid intake
* Patients who have received OPC-41061 in history.
* Participation in any other clinical trial or post-marketing clinical study within 4 weeks prior to informed consent for the present trial
* Female patients who are pregnant, possibly pregnant, or nursing
* Patients otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr., Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (4):
- Japan (4):
  - Kanto, Region
  - Kinki, Region
  - Kyushu, Region
  - Tōhoku, Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-41061 15mg/Day: OPC-41061 (15 mg/day) was orally administered once daily after breakfast on off-dialysis days for 24 weeks.
- OPC-41061 30mg/Day: OPC-41061 (30 mg/day) was orally administered once daily after breakfast on off-dialysis days for 24 weeks.
- Placebo: OPC-41061 placebo was orally administered once daily after breakfast on off-dialysis days for 24 weeks.
Period: Overall Study
Arm/Group | OPC-41061 15mg/Day | OPC-41061 30mg/Day | Placebo
Started | 40 | 40 | 44
Completed | 34 | 36 | 29
Not Completed | 6 | 4 | 15
Not completed — Adverse Event | 3 | 0 | 2
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Met withdrawal criteria | 2 | 2 | 5
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-41061 15mg/Day | OPC-41061 30mg/Day | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 44 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 26 | 22 | 65
  >=65 years | 23 | 14 | 22 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.0) | 60.5 (12.6) | 64.4 (8.7) | 63.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 40 | 56
  Male | 35 | 29 | 4 | 68
Region of Enrollment [Number; unit: participants]
  Japan | 40 | 40 | 44 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Urine Volume
Description: Change in daily urine volume from baseline to the end of the treatment was calculated using descriptive statistics.
Time Frame: Baseline，End of the treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OPC-41061 15mg/Day | OPC-41061 30mg/Day | Placebo
Number analyzed (Participants) | 38 | 38 | 42
mL | 169.2 (422.2) | 111.8 (557.7) | -259.9 (463.8)

2. Secondary Outcome: Change in Total Volume of Fluid Removed by Dialysis Per Week
Description: Change in total volume of fluid removed by dialysis per week from baseline to the end of the treatment was calculated using descriptive statistics.
Time Frame: Baseline，End of the treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OPC-41061 15mg/Day | OPC-41061 30mg/Day | Placebo
Number analyzed (Participants) | 39 | 39 | 43
mL | 485.9 (1979.3) | 375.4 (1721.8) | 1099.5 (2160.5)

ADVERSE EVENTS:
Time Frame: Treatment period
Description: One subject in OPC-41061 15 mg group and one subject in OPC-41061 30 mg group were excluded from all datasets due to the loss of source documents at the site.
Arm/Group | OPC-41061 15mg/Day | OPC-41061 30mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/44
Serious Adverse Events (participants affected / at risk) | 6/39 | 7/39 | 10/44
Other Adverse Events (participants affected / at risk) | 34/39 | 38/39 | 34/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 15mg/Day (N=39) | OPC-41061 30mg/Day (N=39) | Placebo (N=44)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 2
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 1 | 0
Decreased activity (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Occult blood (Investigations) | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 15mg/Day (N=39) | OPC-41061 30mg/Day (N=39) | Placebo (N=44)
Nasopharyngitis (Infections and infestations) | 9 | 14 | 10
Folliculitis (Infections and infestations) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 7 | 3
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 2 | 4
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 4
Vomiting (Gastrointestinal disorders) | 2 | 4 | 1
Blood potassium increased (Investigations) | 2 | 0 | 4
Blood pressure decreased (Investigations) | 3 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Thirst (General disorders) | 4 | 3 | 1
Angina pectoris (Cardiac disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No